CLINICAL TRIAL: NCT03324061
Title: A Phase 1, Randomized, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Fulvestrant (Test vs. Reference) Following Intramuscular Administration to the Gluteal Muscle in Healthy Female Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, and PK of Fulvestrant After IM Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eagle Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EGL-5835-C-1701
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fulvestrant for Injectable Suspension (Experimental): Fulvestrant for Injectable Suspension (500 mg/vial)
  Interventions: Drug: Fulvestrant for Injectable Suspension
- Faslodex (R) (Active Comparator): Faslodex (250 mg/mL)
  Interventions: Drug: Faslodex (Reference)

INTERVENTIONS:
Drug: Fulvestrant for Injectable Suspension — Test drug is administered as a single 5mL intramuscular injection in the right or left dorsogluteal muscle area
  Arms: Fulvestrant for Injectable Suspension
Drug: Faslodex (Reference) — Reference drug is administered as two 5mL intramuscular injections, one in each of the right and left dorsogluteal muscle areas
  Arms: Faslodex (R)

SUMMARY:
Clinical study designed to assess the plasma pharmacokinetic profile and tolerability of Fulvestrant for Injectable Suspension after a single IM dose of Fulvestrant for Injectable Suspension compared to the reference product, Faslodex in healthy female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, parallel group study in healthy female subjects. The study is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of a single dose of Fulvestrant for Injectable Suspension vs. the reference drug, Faslodex, administered in the gluteal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 kg/m2 to 32 kg/m2
* Body weight of at least 50 kg at screening
* Good health as determined by evaluations
* Negative serum pregnancy test
* Subjects who are naturally postmenopausal for at least 12 consecutive months with a follicle-stimulating hormone level at Screening of ≥40 mIU/mL
* Subjects who are peri-menopausal and experiencing at least one of specified symptoms of menopause (eg, hot flashes, mood swings, night sweats, and others)
* Negative urine test for drugs of abuse
* Negative urine test for HIV antibody, HBsAG, and HCV at Screening
* Women of child-bearing potential must agree to consistently practice contraception throughout the duration of the study and continue to do so for 1 year after receiving study drug by one of the following methods: abstinence, condom, diaphragm or cervical cap with spermicide, intrauterine device or male partner had previously undergone a vasectomy as declared in medical history

Exclusion Criteria:

* Recent history (6 months) or current evidence of any clinically significant (uncontrolled) disorder including hepatic, renal, cardiovascular, psychological, pulmonary, metabolic, endocrine, neurologic, infectious, gastrointestinal, hematologic or oncologic disease, or other medical conditions that may interfere with the subject completing the study
* Lab test results outside the normal range at Screening or Day 1 considered clinically significant by the Investigator
* Use of hormonal replacement therapy within 6 months prior to randomization an/or current use of oral contraceptive pill or patch as contraceptive method throughout the study
* Concomitant medication that can affect bleeding
* Recent history (6 months) or presence of an abnormal ECG that, in the opinion of the Investigator, is clinically significant
* Subjects with QTcF interval duration >470 milliseconds
* History of alcoholism or drug addiction within 1 year prior to Day 1
* History of allergy or a known sensitivity to product components of fulvestrant Test and Reference formulations
* Creatinine clearance <60 mL/minute based on the Cockcroft-Gault equation
* Blood donation of 500 mL or more or a significant loss of blood within 56 days prior to Day 1
* Previous exposure to fulvestrant
* Familial relationship with another study participant

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Day 0 through Day 140
  Area under the concentration-time curve(AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian J Hepner, MD, PhD, Study Director — Eagle Pharmaceuticals, Inc.
Locations (12):
- United States (12):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Quotient Sciences, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Clinical Research Consortium, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - New Horizon Clinical Research, Cincinnati, Ohio
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Optimal Research, LLC, Austin, Texas
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No